CLINICAL TRIAL: NCT01879020
Title: A Randomised Double-blind, Placebo-controlled, Ascending-dose, Phase I Study to Determine the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TA-8995 After Multiple Doses in Healthy Adult Male Subjects
Brief Title: Evaluation of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TA-8995 After Multiple Doses in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TA-8995-E02
Record Dates: First submitted 2013-06-04; First posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Dyslipidemia
Keywords: MT-8995; Dyslipidemia; Cholesteryl ester transfer proteins
MeSH Terms: conditions — Dyslipidemias | interventions — TA-8995

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- TA-8995 1 mg (Experimental)
  Interventions: Drug: TA-8995
- TA-8995 2.5 mg (Experimental)
  Interventions: Drug: TA-8995
- TA-8995 5 mg (Experimental)
  Interventions: Drug: TA-8995
- TA-8995 10 mg (Experimental)
  Interventions: Drug: TA-8995
- TA-8995 25 mg (Experimental)
  Interventions: Drug: TA-8995
- Placebo (TA-8995 1mg) (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo (TA-8995 2.5mg) (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo (TA-8995 5mg) (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo (TA-8995 10mg) (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo (TA-8995 25mg) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TA-8995 — Drug: TA-8995 1mg
  Arms: TA-8995 1 mg
Drug: TA-8995 — Drug: TA-8995 2.5mg
  Arms: TA-8995 2.5 mg
Drug: TA-8995 — Drug: TA-8995 5mg
  Arms: TA-8995 5 mg
Drug: TA-8995 — Drug: TA-8995 10mg
  Arms: TA-8995 10 mg
Drug: TA-8995 — Drug: TA-8995 25mg
  Arms: TA-8995 25 mg
Drug: Placebo — Placebo (TA-8995 1mg)
  Arms: Placebo (TA-8995 1mg)
Drug: Placebo — Placebo (TA-8995 2.5mg)
  Arms: Placebo (TA-8995 2.5mg)
Drug: Placebo — Placebo (TA-8995 5mg)
  Arms: Placebo (TA-8995 5mg)
Drug: Placebo — Placebo (TA-8995 10mg)
  Arms: Placebo (TA-8995 10mg)
Drug: Placebo — Placebo (TA-8995 25mg)
  Arms: Placebo (TA-8995 25mg)

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of TA-8995 after multiple doses in healthy adult male subjects

ELIGIBILITY:
Inclusion Criteria:

* Free from any clinically significant illness or disease as determined by their medical history, physical examination, laboratory and other tests and as judged by the Investigator.
* Between 18 - 55 years old.
* Male of Caucasian ethnic origin.
* Body mass index (BMI) in the range of 19 - 33 kg/m² and had a minimum weight of 50 kg. Subjects with a BMI in the range 30.0 - 33.0 kg/m² had to have a waist measurement of ≤ 91 cm.

Exclusion Criteria:

* High density lipoprotein (HDL)-C level of greater or equal to 2.59 mmol/L (≥ 100 mg/dL) at Screening.
* Abnormal Electrocardiogram (ECG) at Screening or Day -1 including a QTc ≥ 430 ms (The QTc-interval was calculated automatically according to Bazett's formula. In the case of results of ≥ 430 ms, QTc was additionally calculated manually using Fridericia's formula which was used as an exclusion criterion).
* Family history of long QT syndrome, hypokalaemia or Torsades de Pointes
* Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease or history of any psychotic illness
* Presence or history of gastro-intestinal, hepatic or renal disease or any other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 336 hours post dose
Laboratory tests (haematology, biochemistry and urinalysis) | 336 hours post dose
Vital signs (supine systolic and diastolic blood pressure, heart rate and body temperature) | 336 hours post dose
Area under the plasma concentration (AUC) versus time curve over the final dosing interval (AUC0-τ, Steady-state) | 7 days post the final dose
The last time point 't' with a concentration Ct ≥ Lower limit quantification (LLQ) (AUC0-t, Steady-state) | 7 days post the final dose

SECONDARY OUTCOMES:
Cholesterol ester transfer protein (CETP) activity (%) | 7 days post the final dose
CETP concentration (mg/mL) | 4 hours after the first and the fibal dose

CONTACTS AND LOCATIONS:
Overall Officials: Werner Weber, MD, Principal Investigator — Momentum Pharma Services GmbH
Locations (1):
- Momentum Pharma Services GmbH, Hamburg, Germany